CLINICAL TRIAL: NCT03033147
Title: Effect of Preoperative, Single-dose Amoxicillin/Clavulanic Acid Combination on Postoperative Endodontic Pain in Patients With Symptomatic Apical Periodontitis: A Double-Blind Randomized Controlled Trial.
Brief Title: Effect of Preoperative Amoxicillin/Clavulanic Acid Combination on Postoperative Endodontic Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nermeen Naser Taleb Moushtaha, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CEBC-CU-2016-12-163
Record Dates: First submitted 2017-01-24; First posted 2017-01-26 (Estimated); Last update posted 2021-06-18 (Actual); Status verified 2021-06

CONDITIONS: Symptomatic Periapical Periodontitis
MeSH Terms: interventions — Amoxicillin; Clavulanic Acid; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amoxicillin/Clavulanate Potassium (Experimental): Amoxicillin/Clavulanate Potassium 875 mg-125 mg orally 30 minutes before root canal treatment
  Interventions: Drug: Amoxicillin/Clavulanate Potassium 875 mg-125 mg oral tablet
- Placebo (Placebo Comparator): placebo 30 minutes before root canal treatment
  Interventions: Drug: Oral placebo

INTERVENTIONS:
Drug: Amoxicillin/Clavulanate Potassium 875 mg-125 mg oral tablet — 2 gm of amoxicillin/ clavulanic acid combination orally 30 minutes before root canal treatment
  Other Names: Augmentin
  Arms: Amoxicillin/Clavulanate Potassium
Drug: Oral placebo — placebo 30 minutes before root canal treatment
  Arms: Placebo

SUMMARY:
The aim of this prospective, randomized, placebo controlled study is to evaluate the effect of a single preoperative dose of amoxicillin/clavulanic acid combination on post-operative pain and swelling in adult patient with symptomatic apical periodontitis.

DETAILED DESCRIPTION:
Medical and dental history will be obtained from all patients participating in this trial. Clinical and radiographic evaluation for each tooth included in this study will be recorded.

Clinical diagnosis of symptomatic apical periodontitis is to be confirmed.

Prior to initiation of root canal treatment, eligible participants will be randomly assigned to one of the following groups: experimental group (receiving 2 gm of amoxicillin/ clavulanic acid orally 30 minutes before the treatment) or control group (receiving a placebo 30 minutes before treatment).

Root canal treatment will then be carried out in a single visit.

Each patient will receive a 7-day diary to record postoperative pain and swelling. In case of pain, the participant will be instructed to take an analgesic. Post-operative pain will be measured as a primary outcome on 11-point scale (NRS) at the following time points: 6, 12, 24, 48, 72 hours and 7 days. The occurrence of swelling will be reported by participant as a secondary outcome.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic apical periodontitis who do not have evidence of spreading infection or systemic involvement.
* Mandibular posterior teeth.
* Patients with non-contributory systemic condition.
* Patients who can understand pain scales and able to sign informed consent.

Exclusion Criteria:

* Patients allergic to penicillin.
* Patients who have a draining sinus tract.
* Retreatment cases.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-10-18 (Actual); Primary Completion 2020-03-15 (Actual); Study Completion 2020-03-15 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | Up to 7 days after endodontic treatment
  Postoperative pain will be measured by a numerical rating scale (NRS).

SECONDARY OUTCOMES:
Swelling | Up to 7 days after endodontic treatment
  The occurrence of Swelling will be measured by a questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Nermeen NT Moushtaha, Postgraduate, Principal Investigator — Cairo University; Suzan AW Amin, PhD, Study Chair — Cairo University; Shaimaa Gawdat, PhD, Study Director — Cairo University
Locations (1):
- Cairo University Faculty of Dentistry, Cairo, Egypt

REFERENCES:
- [Background] Cope A, Francis N, Wood F, Mann MK, Chestnutt IG. Systemic antibiotics for symptomatic apical periodontitis and acute apical abscess in adults. Cochrane Database Syst Rev. 2014 Jun 26;(6):CD010136. doi: 10.1002/14651858.CD010136.pub2. PMID 24967571
- [Background] Akbar I. Efficacy of Prophylactic use of Antibiotics to Avoid Flare up During Root Canal Treatment of Nonvital Teeth: A Randomized Clinical Trial. J Clin Diagn Res. 2015 Mar;9(3):ZC08-11. doi: 10.7860/JCDR/2015/12046.5620. Epub 2015 Mar 1. PMID 25954695
- [Background] Contardo L, Meneguzzi E, Cadenaro M, Di Lenarda R. Clinical evaluation of antibiotic prophylaxis before endodontic treatment of necrotic teeth. Minerva Stomatol. 2005 Mar;54(3):153-60. English, Italian. PMID 15920447
- [Background] Pickenpaugh L, Reader A, Beck M, Meyers WJ, Peterson LJ. Effect of prophylactic amoxicillin on endodontic flare-up in asymptomatic, necrotic teeth. J Endod. 2001 Jan;27(1):53-6. doi: 10.1097/00004770-200101000-00019. PMID 11487166